CLINICAL TRIAL: NCT02253693
Title: Descriptive Pilot Study of Monitoring of Physical Activity in Adult Patients With Haemophilia A Arthropathy by Means of Accelerometry, Image Tests and Physical Condition Parameters. Benefits Associated With That Monitoring"
Brief Title: Exploratory Pilot Study of Physical Activity Monitoring in Adult Patients With Haemophilia A by Means of Accelerometry
Status: Completed | Type: Observational
Sponsor: University of Valencia (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Felipe Querol Fuentes, Full Lecturer, University of Valencia
Other Study IDs: H14-23641
Record Dates: First submitted 2014-09-22; First posted 2014-10-01 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Hemophilia A, Congenital
Keywords: Hemophilia A; Hemophilic arthropathy; Accelerometry
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients with haemophilia: Adult patients with haemophilia A presenting joint disease.

SUMMARY:
Research Question: Does an specific and pre-defined physical exercise prescribed by a specialist provide any benefit on haemophilic arthropathy, the quality of life or the physical condition of patients with haemophilia A and haemophilic arthropathy? Does adherence to physical exercise improve when monitoring patients with an accelerometer? Do compliant patients find higher benefit on haemophilic arthropathy, quality of life or the physical condition than non-compliant patients?

Primary Endpoint: Assess in patients with haemophilia A and haemophilic arthropathy if a prescribed and specific physical exercise monitored by an accelerometer is producing any change in the following domains: progress of haemophilic arthropathy; health-related quality of life; physical condition.

Secondary Endpoints: Evaluate the adherence to physical exercise in patients with haemophilia A and haemophilic arthropathy by means of accelerometry, and asses if compliant patients achieve higher improvement in these 3 domains than non-complaint patients.

DETAILED DESCRIPTION:
Specific details of Treatment/Intervention:

Physical exercises that are part of the specific medical program prescribed for each patient. The exercise program for each patient will depend of the haemophilic arthropathy, the level of physical condition and the preferences of the patient.

Monitoring of physical activity will be made by means of accelerometers. Its use does not alter the daily activities and does not require any change of the patients' individual habits. The assessment of the patients' cardiovascular condition will be made using pulse monitors. Normal examinations in clinical practice will be revised as well as those specific to each patient reference health centre, muscle strength and joint use testing which will be validated with force measurement devices. Assess by means of an ultrasound system the baseline situation of the joints used for daily activities for injury control. Determine the likelihood of fracture and assess the bone quality by means of densitometry. Thermal cameras will allow to analyse the characteristics of Joint inflammation. It may be suitable for bleeding evolution control. Measurements given by densitometers will allows to determine the state of bones of the participants in the study (osteoporosis measurement). Number of bleeding events/hemarthrosis during the period of study. Determine the activity of hemarthros/synovitis using thermal images.

ELIGIBILITY:
Inclusion Criteria:

* Male patients over 18
* Patients diagnosed with haemophilia A and under prophylaxis treatment with the same FVIII for 2 years prior to the inclusion in the study.
* Patients with haemophilic arthropathy in, at least, one of the four load-bearing joints (knees and ankles), according to clinical and/or radiographic criteria (at least 3 in the Gilbert scale and /or at least 3 in the Pettersson scale) and/or Chronic synovitis evidenced by ultrasound.
* Patients with signed informed consent.

Exclusion Criteria:

* Patients who have developed an inhibitor antibody (≥5 Bethesda units), at the moment of the inclusion in the study.
* Development of inhibitors
* Modification, during follow-up, of FVIII with which the patient started the study.
* The patient decides to withdraw voluntarily from the study.
* Major orthopaedic surgery

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with haemophilia A presenting joint disease (haemophilic arthropathy) and who are under prophylaxis treatment with FVIII
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the physiotherapy treatment compliance. Parameters: Intensity, duration, type of exercise and % of compliance. | After 6, 12, 18 and 24 months.
  Level of treatment compliance assessed by the intensity (counts/min), duration (m) and type of exercise measured with triaxial accelerometer.

SECONDARY OUTCOMES:
Age (years). | In month 0, and month 24.
  Age of patient.
Weight (Kg). | In month 0, and month 24.
  Weight of patient.
Biochemistry and haemogram tests. The parameters to be reported are: Leukocyte (mil/mm3), Lymphocyte (mil/mm3), Haemoglobin (g/dl), Glucose (mg/dl), Total, HDL and LDL cholesterol (mg/dl), Triglyceride (mg/dl) and Creatine phosphokinase (CPK) (UI/L). | In Baseline and after 6, 12, 18 and 24 months.
Prophylactic treatment with Factor VIII. Parameters: Trough levels of FVIII in blood (% FVIII) and type of FVIII and dose (UI/ week). | In Baseline and after 6, 12, 18 and 24 months.
Body composition of patient. Parameters: BMI (Kg/m^2) and % of body fat. | In Baseline and after 6, 12, 18 and 24 months.
Cardiovascular condition. Parameters: Beats/minute and distance covered (metres). | In Baseline and after 6, 12, 18 and 24 months.
  Beats/minute measured with a pulse monitor and distance covered in Six-minute walk test (6MWT).
Blood pressure (mmHg). | In Baseline and after 6, 12, 18 and 24 months.
  Measured with Cuff- stethoscope; Manometer; manual meter.
Muscle strength in kilos (peak force and time to reach peak force). | In Baseline and after 6, 12, 18 and 24 months.
  Measured with Lafayette device.
State of joints and injury control (HJHS 2.1. score). | In Baseline and after 6, 12, 18 and 24 months.
  Evaluated by ultrasound system.
Joint inflammation. Parameters: Thermal imaging (ºC) and joint perimeter (cm). | In Baseline and after 6, 12, 18 and 24 months.
  Measured with thermal camera and tape measure.
Bone density. Parameter: Bone Quality Index (BQI). | In Baseline and in month 24.
  Densitometry.
Bleeding/ hemarthrosis. Parameter: Bleeding Rate (BR). | In Baseline and after 6, 12, 18 and 24 months.
  Registered in patient's diary.
Health-related quality of life. Parameters: General questionnaire (EQ-5D EuroQoL) and specific questionnaire (A36 Hemophilia QoL). | In Baseline and in 12 and 24 month.

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Querol-Fuentes, Principal Investigator — University of Valencia
Locations (2):
- Spain (2):
  - University of Valencia, Valencia
  - Hospital Universitari i Politècnic La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodríguez-Merchan EC, Goddard NJ, Lee CA, editors. Musculoskeletal Aspects of Haemophilia. Oxford: Blackwell Sciencie Ltd; 2000.
- [Background] Gonzalez LM, Peiro-Velert C, Devis-Devis J, Valencia-Peris A, Perez-Gimeno E, Perez-Alenda S, Querol F. Comparison of physical activity and sedentary behaviours between young haemophilia A patients and healthy adolescents. Haemophilia. 2011 Jul;17(4):676-82. doi: 10.1111/j.1365-2516.2010.02469.x. Epub 2011 Feb 7. PMID 21299746
- [Background] Hendelman D, Miller K, Baggett C, Debold E, Freedson P. Validity of accelerometry for the assessment of moderate intensity physical activity in the field. Med Sci Sports Exerc. 2000 Sep;32(9 Suppl):S442-9. doi: 10.1097/00005768-200009001-00002. PMID 10993413